CLINICAL TRIAL: NCT05760833
Title: Pulmonary Vein Isolation or Atrioventricular Node Ablation in Patients With Heart Failure and Symptomatic Atrial Fibrillation Diminishing CRT Response (PULVERISE-AF-CRT): a Randomized Study
Brief Title: Ablation in Patients With HF and Symptomatic AF: PULVERISE-AF-CRT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No inclusion
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PULVERISE-AF-CRT
Record Dates: First submitted 2022-12-22; First posted 2023-03-08 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2023-03

CONDITIONS: Atrial Fibrillation; Heart Failure
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulmonary vein isolation (Active Comparator): Ablation of the pulmonary veins.
  Interventions: Procedure: Ablation
- atrioventricular node ablation. (Active Comparator): Ablation of the atrioventricular node.
  Interventions: Procedure: Ablation

INTERVENTIONS:
Procedure: Ablation — Ablation of either the pulmonary veins or the atrioventricular node

SUMMARY:
Pulmonary vein isolation (PVI) is currently the cornerstone non pharmacological therapy for drug-refractory atrial fibrillation (AF). Where rhythm control has been shown to be inferior as compared to rate control in older trials. New data suggest that for patients with heart failure and AF PVI may improve prognosis (mortality) as compared to medical rate or rhythm control. Whether optimal rate control as can be achieved with atrioventricular node ablation is comparable with regard to all-cause mortality of heart failure hospitalization to PVI in patients with heart failure and AF is unknown.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a cardiac resynchronization therapy device (CRT-D or CRT-P) and optimal medical therapy according to current guidelines.
* Patients with paroxysmal or persistent AF, having AF or HF related symptoms.
* Patient with paroxysmal AF should have >25% burden or inadequate biventricular pacing (<95%) based on device counters.
* The patient is willing and able to comply with the protocol and has provided written informed consent.
* Age ≥ 18 years

Exclusion Criteria:

* Documented left atrial diameter > 6 cm (parasternal long axis).
* Longstanding persistent AF longer than 2 years.
* Contraindication to chronic anticoagulation therapy or heparin
* Previous left heart ablation procedure for AF
* Acute coronary syndrome, cardiac surgery, angioplasty or stroke within 2 months prior to enrolment
* Untreated hypothyroidism or hyperthyroidism
* Enrolment in another investigational drug or device study.
* Woman currently pregnant or breastfeeding or not using reliable contraceptive measures during fertility age.
* Mental or physical inability to participate in the study.
* Listed for heart transplant.
* Cardiac assist device implanted.
* Planned cardiovascular intervention.
* Life expectancy ≤ 12 months.
* Uncontrolled hypertension.
* Requirement for dialysis due to terminal renal failure.
* Participation in another telemonitoring concept

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2024-04-08 (Actual)

PRIMARY OUTCOMES:
All-cause death. | 1 year
  Occurence of all-cause death.
cardiovascular hospitalization. | 1 year
  Occurence of cardiovascular hospitalization (heart failure or stroke).
Quality of life | 1 year
  Change in quality of life (using the Kansas City Cardiomyopathy Questionnaire (KCCQ)).

SECONDARY OUTCOMES:
Death from any cause | 1 year
  Occurence of death from any cause.
Unplanned hospitalization | 1 year
  Occurence of unplanned hospitalization related to heart failure.
death from cardiovascular disease | 1 year
  Occurence of death from cardiovascular disease.
cerebrovascular accident. | 1 year
  Occurence of stroke.
unplanned hospitalization for cardiovascular disease | 1 year
  Any unplanned hospitalization for cardiovascular disease.
Any hospitaliation | 1 year
  Any hospitalization for non-cardiovascular disease.
changes in the Kansas city cardiomyopathy questionnaire | 1 year
  Changes in quality of life (any)
procedure related adverse events | 1 year
  Occurence of procedure related adverse events.
atrial fibrillation-free intervals were assessed. | 1 year
  Assessment of AF free intervals.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided